CLINICAL TRIAL: NCT02768480
Title: Evaluation of the Effectiveness of Phone Calls Intervention (TelessaúdeRS) on Diabetic Patients After Ambulatory Discharge of a Tertiary Care Center: A Randomized Clinical Trial
Brief Title: Effectiveness of Phone Calls Intervention on Diabetic Patients After Ambulatory Discharge of a Tertiary Care Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 150503
Record Dates: First submitted 2016-04-29; First posted 2016-05-11 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; phone calls; glycemic control
MeSH Terms: conditions — Diabetes Mellitus | interventions — Primary Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Primary Care (Active Comparator): Patients will be followed by primary care team exclusively.
  Interventions: Other: Primary Care
- Phone Calls Support and Primary Care (Experimental): Patients will be followed by primary care team and supported by periodic nurse phone calls.
  Interventions: Other: Phone Calls Support and Primary Care

INTERVENTIONS:
Other: Primary Care — Patients will be followed by primary care team according to the usual health system routine.
  Arms: Primary Care
Other: Phone Calls Support and Primary Care — Patients in intervention group will receive periodic phone calls (every three months) and will have a toll-free number to resolve questions about the disease management. The phone-calls will be performed by trained nurses and will follow a structured format. Nurses will address some topics: patient's treatment adherence, technique of insulin administration, disease understanding, hypoglycaemia management, healthy diet, smoke cessation and foot care.
  Arms: Phone Calls Support and Primary Care

SUMMARY:
The study is a randomized clinical trial, controlled, open label that aimed to compare two groups after discharge of a tertiary care: type 2 diabetes patients followed exclusively by primary care (control group) and patients followed by primary care and supported by phone calls (intervention group).

DETAILED DESCRIPTION:
The investigators designed a randomized controlled trial. Patients with stable and controlled type 2 diabetes, and considered to be eligible to discharge from specialized care to primary care will be included. Patients with severe neuropathy, not controlled ischemic heart disease and nephropathy stage IV/V will be excluded. Enrolled patients will be randomized in two groups: follow-up supported by periodic nurse phone calls plus primary care (intervention group) or followed by primary care team (control group). The intervention group will receive regular telephone calls (every 3 months for 1 year) and will have a toll-free number to resolve questions about the disease management. Main outcome is the glycemic control between groups after 1 year of follow-up. Secondary outcomes include: rate of hypoglycaemia, blood pressure control,emergency visits, nephropathy progression and death.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes;
* Patients who met discharges criteria according to endocrinology team;
* Patients with HbA1C < 8%.

Exclusion Criteria:

* Patients with stage IV or V nephropathy;
* Patients with not controlled Ischemic heart disease;
* Patients with severe autonomous or peripheral neuropathy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2015-06; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Glycemic Control | 1 year
  Evaluation after 1 year of discharge with HbA1c

SECONDARY OUTCOMES:
Visits to the doctor, nurse, nutritionist, psychologist | 1 year
  Evaluation after 1 year of discharge with a structured questionnaire
Rate of referring to tertiary care | 1 year
  Evaluation after 1 year of discharge with a structured questionnaire
Care satisfaction with diabetes treatment | 1 year
  Evaluation after 1 year of discharge with a structured questionnaire
Emergency visits because of diabetes acute complications | 1 year
  Evaluation after 1 year of discharge with a structured questionnaire
Hypoglycaemic rate | 1 year
  Evaluation after 1 year of discharge with a structured questionnaire
Treatment adherence | 1 year
  Evaluation after 1 year of discharge with the Brief Medication Questionnaire
Lipid control | 1 year
  Evaluation after 1 year of discharge with blood lipid levels
Antiplatelet therapy/ statin use | 1 year
  Evaluation after 1 year of discharge with a structured questionnaire
Nephropathy emergence or worsening | 1 year
  Evaluation after 1 year of discharge with microalbuminuria and blood creatinine measurement
Retinopathy emergence or worsening | 1 year
  Evaluation after 1 year of discharge with retinography and ophthalmologist advice if is necessary.
Major cardiovascular events | 1 year
  Evaluation after 1 year of discharge with a structured questionnaire
Death | 1 year
  Evaluation after 1 year of discharge with telephone contact and active search

OTHER OUTCOMES:
Blood Pressure | 1 year
  Evaluation after 1 year of discharge with blood pressure measurement

CONTACTS AND LOCATIONS:
Overall Officials: Sandra P Silveiro, MD, Study Director — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moreira AM, Rados DV, de Farias CB, Coelli S, de Almeida Faller L, Dos Santos LF, Matzenbacher AM, Katz N, Harzeim E, Silveiro SP. Effects of nurse tele support via telephone calls on transition between specialized and primary care in type 2 diabetes mellitus patients: a CONSORT-compliant randomized clinical trial. Endocrine. 2025 Mar;87(3):978-986. doi: 10.1007/s12020-024-04095-6. Epub 2024 Nov 29. PMID 39614069
- [Derived] Moreira AM, Marobin R, Rados DV, de Farias CB, Coelli S, Bernardi BL, Faller LA, Dos Santos LF, Matzenbacher AM, Katz N, Harzheim E, Silveiro SP; TelessaudeRS. Effects of nurse telesupport on transition between specialized and primary care in diabetic patients: study protocol for a randomized controlled trial. Trials. 2017 May 18;18(1):222. doi: 10.1186/s13063-017-1954-z. PMID 28521796